CLINICAL TRIAL: NCT07291011
Title: A Pilot Study of Mindfulness-Based Stress Reduction (MBSR) in Patients With Cancer Experiencing Stress Who Live in Underserved and Rural Regions of Minnesota
Brief Title: A Mindfulness-Based Stress Reduction Program for Improving Mental Health Outcomes for Underserved Cancer Patients in Minnesota
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 24-013451; NCI-2025-08924 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 24-013451 (Other: Mayo Clinic Institutional Review Board)
Record Dates: First submitted 2025-12-05; First posted 2025-12-18 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Hematopoietic and Lymphatic System Neoplasm; Malignant Solid Neoplasm
MeSH Terms: interventions — Mindfulness; Mindfulness-Based Stress Reduction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Supportive care (MBSR) (Experimental): Patients participate in MBSR sessions weekly for 8 weeks.
  Interventions: Other: Electronic Health Record Review; Behavioral: Mindfulness Relaxation; Other: Questionnaire Administration

INTERVENTIONS:
Other: Electronic Health Record Review — Ancillary studies
Behavioral: Mindfulness Relaxation — Receive MBSR intervention
  Other Names: MBSR; Mindful Meditation; Mindfulness Meditation; Mindfulness-Based Stress Reduction
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This clinical trial evaluates whether a virtual stress reduction program that uses mindfulness-based stress reduction (MBSR) techniques works to improve mental health outcomes in cancer patients living in underserved/rural regions of Minnesota. 80% of Minnesota counties are considered mental health care shortage areas. This shortage disproportionately impacts Minnesotans living in underserved and rural regions as they have to travel further for mental health care services. Interventions that provide patients with mental health resources from the comfort of their own home help to reduce barriers that limit access to mental health care. MBSR courses can help patients control their responses to stressful events, reduce the impact of chronic stress, develop more effective ways to cope with medical/psychological conditions, and increase overall sense of well-being. MBSR courses may serve as a way to bridge the gap between mental health care and patients with cancer living in underserved/rural regions of Minnesota.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a history of cancer, or currently have cancer
* Patients reporting > 4/10 emotional distress on a 0-10 scale within the past two weeks
* Have a computer or smartphone
* Willing to complete questionnaires

Exclusion Criteria:

* Non-English-speaking patients
* Life expectancy < 12 months
* Active psychiatric disease

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-11-05 (Actual); Primary Completion 2027-11-15 (Estimated); Study Completion 2029-11-15 (Estimated)

PRIMARY OUTCOMES:
Completion Rate | Up to 10 weeks
  Assessed by the number of participants who complete the virtual stress reduction program (MBSR) program
Change in Stress | Baseline, at completion of 8-week course, 3 months, 6 months
  Assessed using the 10-item Perceived Stress Scale (PSS), which measures global perceived stress experienced by the participant over the preceding 30 days. The PSS consists of 10 questions assessing how often the participant felt or thought a certain way during the past month. Possible answers include: 0 - never; 1 - almost never; 2 - sometimes; 3 - fairly often, and 4 - very often. Possible scores range from 0 to 40, with lower scores indicating a better outcome (less stress).
Change in Anxiety | Baseline, at completion of 8-week course, 3 months, 6 months
  Assessed using the General Anxiety Disorder 7-item (GAD-7) scale. The GAD-7 consists of 7 questions answered on a scale of 0-3 where 0=not at all, 1=several days, 2=more than half the days, and 3=nearly every days. The total score ranges from 0 to 21 where 0 indicates no anxiety, 1-4 indicates minimal anxiety, 5-9 indicates mild anxiety, 10-14 indicates moderate anxiety, and 15-21 indicates severe anxiety.
Change in Mindfulness | Baseline, at completion of 8-week course, 3 months, 6 months
  Assessed using the Mindful Attention Awareness Scale (MAAS), a 15-item scale designed to assess a core characteristic of dispositional mindfulness (open or receptive awareness of and attention to what is taking place in the present). The MAAS consists of 15 statements about everyday experience, with each item answered on a scale ranging from 1 (almost always) to 6 (almost never) to indicate how frequently or infrequently participants have each experience. The MAAS is scored by computing a mean (average) of all 15 items. Higher scores reflect higher levels of dispositional mindfulness.
Barriers to completion of the course | 10 weeks post course enrollment
  Assessed using a study-specific questionnaire. Responses will be evaluated and reported descriptively.

CONTACTS AND LOCATIONS:
Overall Officials: Stacy D D'Andre, Principal Investigator — Mayo Clinic in Rochester
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States